CLINICAL TRIAL: NCT00783835
Title: A Multicenter Open Trial to Evaluate the Effectiveness and Quality of Life in Adults With Attention Deficit /Hyperactivity Disorder (ADHD) Treated With Long Acting Methylphenidate (CONCERTA)
Brief Title: Study to Evaluate the Efficacy and Quality of Life of Long-Acting Methylphenidate in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013999; 42603ATT4053; NCT00783835
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2013-07-23 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; Methylphenidate; Concerta; CONQoL
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylphenidate (Experimental)
  Interventions: Drug: Long-Acting Methylphenidate

INTERVENTIONS:
Drug: Long-Acting Methylphenidate — Long-Acting Methylphenidate within the range of 18, 36, 54 and 76 milligram will be orally administered once daily up to Day 56.
  Other Names: Concerta

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and to assess the impact of the treatment on quality of life of long-acting methylphenidate in adult participants with Attention Deficit Hyperactivity Disorder (ADHD). ADHD is a clinical condition beginning in childhood and is characterized by inadequate levels of attention, hyperactivity and impulsiveness.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (when more than one hospital or medical school team work on a medical research study), single arm study of multiple doses of long-acting methylphenidate in participants with ADHD. The study will consist of 2 phases; a screening phase and a treatment phase. The duration of participation in the study for an individual participant will be up to 12 weeks. Participants will be given 18 milligram (mg) of long-acting methylphenidate daily in the morning and titrated up (slow increase in drug dosage guided by participant's responses) to 36 mg per day (mg/day) on Day 8. Depending on response, tolerability and clinician's judgment, the dose could be escalated to the next dose level of 54 mg/day on Day 28 to a maximum of 72 mg/day on Day 56, until each participant achieved optimal dose. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Attention Deficient Hyperactivity Disorder (ADHD) according to the Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition (DSM-IV), obtained via interview with an adapted version of the Kiddie-Schedule of Affective Disorders and Schizophrenia-Epidemiologic Version (K-SADS E) module for ADHD
* Described chronic course of ADHD symptomatology from childhood to adulthood, with some symptoms present before age 7 years, which continue to meet DSM-IV criteria at the time of assessment. ADHD is not diagnosed if the symptoms are better accounted for by another psychiatric disorder [e.g. mood disorder (especially bipolar disorder), anxiety disorder, psychotic disorder, personality disorder]
* Clinical Global Impression-Severity (CGI-Severity) baseline score greater than or equal to (>=) 4 (at least moderate severity)
* Female participants must be postmenopausal (after the time in life when a woman stops having a menstrual period) for at least 1year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives[compounds, usually hormonal, taken orally in order to block ovulation and prevent the occurrence of pregnancy], contraceptive injections [chemical substances that prevent or reduce the probability of pregnancy], intrauterine device [contraceptive devices placed high in the uterine fundus], double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study; have a negative urine pregnancy test at baseline
* Participant agrees to take only the supplied study drug as treatment for ADHD during the study

Exclusion Criteria

* Participant having allergy or hypersensitivity to methylphenidate
* Participants who are non-responder to methylphenidate in adequate doses (i.e., 0.8 - 1.0 milligram per kilogram [mg/kg])
* Participant treated with any methylphenidate or amphetamine containing medication within 4 weeks of the screening visit
* Participant having Hamilton's Depression Scale, suicide item higher than 2
* Participant having any psychiatric condition including the following, but not limited to: acute mood disorder (disorders that have a disturbance in mood as their main feature), schizophrenia (a mixed psychiatric disorder relating to a complex psychotic state that has features of both schizophrenia and a mood disorder such as bipolar disorder), bipolar disorder I (disorder marked by severe mood swings (manic or major depressive episodes) and a tendency to remission [when a medical problem gets better or goes away at least for a while] and recurrence [happen again]), obsessive compulsive disorder (OCD) (an anxiety disorder characterized by recurrent, persistent obsessions or compulsions, anti-social personality disorder ( personality disorder whose essential feature is a pervasive pattern of disregard for, and violation of, the rights of others that begins in childhood or early adolescence and continues into adulthood)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (5):
- Brazil (5):
  - Belo Horizonte
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - São Paulo

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylphenidate: Oral long acting methylphenidate tablets were administered daily at a starting dose of 18 milligram (mg) and slowly increased to 36 mg on Day 8. Depending on response, tolerability and clinician's discretion, the dose could be increased to 54 mg on Day 28 to a maximum of 72 mg per day on Day 56, until each participant achieved optimal dose.
Period: Overall Study
Arm/Group | Methylphenidate
Started | 60
Completed | 50
Not Completed | 10
Not completed — Adverse Event | 3
Not completed — Medical Criteria | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Participant not Adherent | 3

BASELINE CHARACTERISTICS:
Arm/Group | Methylphenidate
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Adult Attention Deficit Hyperactivity Disorder (ADHD) Self-Report Scale (ASRS) Total Score at Week 4
Description: Adult ASRS assesses 18 core ADHD symptoms corresponding to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic symptoms for adult participant based on the participant's own rating for each of the symptoms using a 4 point scale (0=none, 1=mild, 2=moderate, 3=severe). If a single item is missing the score is imputed and if more than one item is missing, the total score is treated as missing. The ASRS total score is derived by summing the score assigned to each of the 18 symptoms (low=0, high=54, a higher score signifies a greater severity of symptoms).
Time Frame: Baseline and Week 4
Population: Intent to treat efficacy evaluation (ITTe) included all participants who received at least 1 dose of study medication and provided at least 1 post-baseline measure of effectiveness.
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale
  Baseline | 52.6 (1.6)
  Change at Week 4 | -10.9 (1.6)

2. Primary Outcome: Change From Baseline in Adult Attention Deficit Hyperactivity Disorder (ADHD) Self-Report Scale (ASRS) Total Score at Week 8
Description: Adult ASRS assesses 18 core ADHD symptoms corresponding to DSM-IV diagnostic symptoms for adult participant based on the participant's own rating for each of the symptoms using a 4 point scale (0=none, 1=mild, 2=moderate, 3=severe). If a single item is missing the score is imputed and if more than one item is missing, the total score is treated as missing. The ASRS total score is derived by summing the score assigned to each of the 18 symptoms (low=0, high=54, a higher score signifies a greater severity of symptoms).
Time Frame: Baseline and Week 8
Population: ITTe included all participants who received at least 1 dose of study medication and provided at least 1 post-baseline measure of effectiveness.
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale | -16.2 (1.6)

3. Primary Outcome: Change From Baseline in Adult Attention Deficit Hyperactivity Disorder (ADHD) Self-Report Scale (ASRS) Total Score at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale | -20.6 (1.7)

4. Primary Outcome: Change From Baseline in Adult ADHD Quality of Life (AAQoL) Scale Score at Week 4
Description: The AAQoL is a validated 29-item scale consisting of 4 subscales:life productivity (11 items), psychological health (6 items), life outlook (7 items) and relationships (5 items). Participants rate each item on a 5-point Likert - like scale ranging from 1 (not at all/never) to 5 (extremely/very often). These scores are then transformed to a 0-100 point scale, higher scores indicating better quality of life. Total score=average of individual 29 item scores (range= 0-100, where higher total score indicates better quality of life). Change from baseline in total score for AAQoL is reported.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale
  Baseline | 39.6 (2.1)
  Change at Week 4 | 19.4 (2.3)

5. Primary Outcome: Change From Baseline in Adult ADHD Quality of Life (AAQoL) Scale Score at Week 12
Description: as for outcome 4
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale | 21.9 (2.3)

6. Secondary Outcome: Change From Screening in Clinical Global Impression-Severity of Illness (CGI-S) Score at Weeks 4, 8 and 12
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 = "Normal, not at all ill" and a rating of 7 = "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Screening (Week -2), 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale
  Screening (Week -2) | 4.6 (0.1)
  Change at Week 4 | -1.0 (0.1)
  Change at Week 8 | -1.3 (0.1)
  Change at Week 12 | -1.7 (0.1)

7. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse).
Time Frame: Week 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale
  Week 4 | 2.7 (0.1)
  Week 8 | 2.4 (0.1)
  Week 12 | 2.2 (0.1)

8. Secondary Outcome: Change From Baseline in the State-Trait Anxiety Inventory (STAI) Scale
Description: The STAI scale consists of total 40 items on separate scales measuring state (20 items) and trait (20 items) anxiety. The participant reports how they feel right now at this moment for state anxiety and how they generally feel for trait anxiety. The state items are scored as: 1 (not at all), 2 (somewhat true), 3 (moderately true), 4 (very true). The trait items are scored as: 1 (almost never), 2 (sometimes), 3 (often), 4 (almost always). The total scores range from 4-80 for each scale. Higher scores indicate more impaired participants.
Time Frame: Baseline, Week 4, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale
  State Anxiety Score: Baseline | 50.4 (1.4)
  Trait Anxiety Score: Baseline | 52.7 (1.5)
  State Anxiety Score: Change at Week 4 | -6.1 (1.2)
  Trait Anxiety Score: Change at Week 4 | -8.4 (1.3)
  State Anxiety Score: Change at Week 8 | -7.8 (1.3)
  Trait Anxiety Score: Change at Week 8 | -8.4 (1.3)
  State Anxiety Score: Change at Week 12 | -9.4 (1.3)
  Trait Anxiety Score: Change at Week 12 | -10.7 (1.3)

9. Secondary Outcome: Change From Screening in the Hamilton Depression Rating (HAM-D) Scale Score at Week 4 and 12
Description: It is a 21-item clinician-rated scale that evaluates depressed mood as well as the vegetative and cognitive symptoms of depression. 11 items are scored on a 3 point scale (0=none/absent to 2=most severe), 2 items are scored on a 4 point scale (0=none/absent to 3=most severe) and 8 items are scored on a 5 point scale (0=none/absent to 4=most severe). The individual items are summed to yield the HAM-D total score that ranges from 0-60, where higher scores indicate worsening.
Time Frame: Screening (Week -2), 4 and 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Unit on a scale
Arm/Group | Methylphenidate
Number analyzed (Participants) | 58
Unit on a scale
  Screening (Week -2) | 5.9 (0.6)
  Change at Week 4 | -2.8 (0.6)
  Change at Week12 | -3.3 (0.6)

ADVERSE EVENTS:
Time Frame: Baseline up to end of study.
Description: An adverse event may be an undesirable and unintended sign (including an abnormal measurement), symptom or disease which is related to the study drug in terms of time regardless of the existence of a causal relationship with the study drug.
Arm/Group | Methylphenidate
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 48/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methylphenidate (N=60)
Tachycardia (Cardiac disorders) | 9
Dry mouth (Gastrointestinal disorders) | 14
Irritability (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 19
Nausea (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 18
Somnolence (Nervous system disorders) | 3
Affect lability (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 6
Initial insomnia (Nervous system disorders) | 6
Insomnia (Nervous system disorders) | 6
Libido decreased (Nervous system disorders) | 4
Nervousness (Nervous system disorders) | 3
Sleep disorder (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo.